CLINICAL TRIAL: NCT03654482
Title: Pilot Study of SuperSeton Placement in Patients With Perianal Fistulas
Brief Title: SuperSeton Pilot Studie
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Proctos Kliniek (Other); MediShield B.V. (Unknown); Delft University of Technology (Other)
Responsible Party: Principal Investigator, Prof. dr. W.A. Bemelman, PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016_018
Record Dates: First submitted 2018-08-15; First posted 2018-08-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Perianal Fistula; Perianal Crohn Disease
Keywords: Knotless seton; Quality of life; Perianal Disease Activity Index

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SuperSeton arm (Experimental)
  Interventions: Device: SuperSeton

INTERVENTIONS:
Device: SuperSeton — The SuperSeton will be placed at the outpatient clinic in patients that already have a seton in situ. This seton will then be exchanged by the SuperSeton. In case patients do not have a seton in situ, the SuperSeton can be placed at the operating theatre in day care setting instead of a regular seton.

SUMMARY:
Rationale: Perianal fistulas are a common incapacitating problem. Many patients are treated by seton drainage to prevent recurrent abscess formation. Nowadays, vessel loops or sutures are used for drainage. The knot of these seton drains can cause complaints of pain or tenderness if it presses against the external opening of the fistula or even slides in to the fistula tract. Medishield B.V. designed a knotless seton drain, the SuperSeton. This could decrease the pain complaints caused by the knot.

Objective: The aim of this study is to determine the feasibility of SuperSeton placement in patients with perianal fistulas.

Study design: The design of the study is a feasibility study.

Study population: Patients (≥ 18 years) with perianal fistulas (ever) treated with a knotted seton are eligible.

Intervention: The SuperSeton will be placed at the outpatient clinic in patients that already have a seton in situ. This seton will then be exchanged by the SuperSeton. In case patients do not have a seton in situ, the SuperSeton can be placed at the operating theatre in day care setting instead of a regular seton.

Main study parameters/endpoints: The primary outcome is seton failure (loosening of the seton). Secondary outcomes are time of procedure, complications and quality of life measured by the PDAI ('Perianal Disease Activity Index').

Nature and extent of the burden and risks associated with participation: The SuperSeton will be placed in patients with perianal fistulas (ever) treated with a conventional knotted seton. There are no additional risks involved. The seton will be placed at the outpatient clinic in patients with a seton in situ, or at the operating theatre in day care setting in patients with a perianal abscess without a seton. The material that is used for the Setons is of medical grade polyurethane, this is the same material of catheters that are already used in clinical practice (instech BTPU 027). The Setons including the insert (BTPU) are supplied sterile (Synergy Health). Sample size calculation: A group of 60 patients will be included to determine feasibility of the SuperSeton. The proposed treatment protocol is considered feasible if at least 70% of the SuperSetons stay in place.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* Written informed consent
* Perianal fistula with a seton in situ or a recurrent perianal fistula for which a new seton will be placed

Exclusion Criteria:

* Patients with a pacemaker or an ICD in situ
* Rectovaginal fistula
* Patients with a stoma
* Life expectancy < 2 years
* The inability of reading/understanding and filling in the questionnaires
* Dementia or altered mental status that would prohibit the understanding and giving of informed consent
* Participation in another trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-08-10 (Actual); Primary Completion 2018-07-04 (Actual); Study Completion 2018-07-04 (Actual)

PRIMARY OUTCOMES:
Seton failure | 3 months
  Loosening of the seton

SECONDARY OUTCOMES:
Perianal Disease Activity Index score | 3 months
  The PDAI is the gold standard for evaluating the severity of perianal disease. It includes five items: discharge, pain, restriction of sexual activity, type of perianal disease, and degree of induration. Each category is graded on a five-point Likert scale ranging from no symptoms to severe symptoms. The sum of the five subscores represents the total PDAI score.
Procedure time | 3 months
Number of participants experiencing complications | 3 months
  Number of participants experiencing peri-operative complications, an increase in perianal pain complains, and perianal abscesses.
Number of participants requiring surgical re-interventions | 3 months

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2017-05-16): https://cdn.clinicaltrials.gov/large-docs/82/NCT03654482/Prot_000.pdf